CLINICAL TRIAL: NCT05164133
Title: A Phase Ib, Single-Arm, Open-Label Study Evaluating the Pharmacokinetics, Pharmacodynamics, and Safety of Tocilizumab in Pediatric Patients Hospitalized With COVID-19
Brief Title: A Study Evaluating Tocilizumab in Pediatric Patients Hospitalized With COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA43811
Record Dates: First submitted 2021-12-16; First posted 2021-12-20 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): Participants who are hospitalized with COVID-19 and who are receiving systemic corticosteroids and require supplemental oxygen or mechanical ventilation will receive a single dose of TCZ on Day 1, with the option to receive a second dose 8-24 hours later if clinically indicated.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants will receive intravenous (IV) tocilizumab

SUMMARY:
This is a single-arm, open-label study to assess the pharmacokinetics, pharmacodynamics, safety, and exploratory efficacy of tocilizumab (TCZ) for the treatment of pediatric patients from birth to less than 18 years old hospitalized with COVID-19 and who are receiving systemic corticosteroids and require supplemental oxygen or mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with COVID-19 confirmed per a positive PCR of any specimen (e.g., respiratory, blood, urine, stool, or other bodily fluid) and evidenced by chest x-ray or CT scan
* Receiving systemic corticosteroids at baseline
* Oxygen saturation < 93% on room air, or requiring supplemental oxygen, non-invasive or invasive mechanical ventilation, or extracorporeal membrane oxygenation (ECMO) to maintain oxygen saturation > 92% at screening and baseline

Exclusion Criteria:

* Gestational age < 37 weeks
* Known severe allergic reactions to TCZ or other monoclonal antibodies
* Active tuberculosis infection
* Uncontrolled active bacterial, fungal, viral, or other infection (besides COVID-19)
* Diagnosis or suspected diagnosis of multisystem inflammatory syndrome in children (MIS-C)
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 48 hours, irrespective of the provision of treatments
* Have received oral anti-rejection or immunomodulatory drugs (including TCZ) within the past 3 months prior to enrollment
* Treatment with an investigational drug within 5 drug-elimination half-lives or 30 days, whichever is longer, of enrollment (except for anti-SARS-CoV-2 antibodies or directly-acting antivirals)
* Participating in another interventional drug clinical trial (except for anti-SARS-CoV-2 antibodies or directly-acting antivirals)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Serum concentration of TCZ | Through Day 28
Maximum serum concentration (Cmax) of TCZ | Through Day 28
Area under the curve from Days 0-28 (AUC days 0-28) of TCZ | Days 0-28
Serum concentration on Day 28 (C day 28) of TCZ | Day 28
Clearance (CL) of TCZ | Through Day 28
Volume of distribution of TCZ | Through Day 28

SECONDARY OUTCOMES:
Duration of 90% saturation of sIL-6R | Through Day 28
Concentration of IL-6 | Through Day 60
Concentration of sIL-6R | Through Day 60
Concentration of C-reactive protein (CRP) | Through Day 60
Percentage of participants with adverse events | Up to 60 days
Percentage of participants with severe adverse events | Up to 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- United States (7):
  - Reagan UCLA Medical Center, Los Angeles, California
  - The University of Chicago, Chicago, Illinois
  - Central Michigan University College of Medicine, Mount Pleasant, Michigan
  - Feinstein Institute for Medical Research, Manhasset, New York
  - University Hospitals Cleveland Medical Center, Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - UT Physicians - Pediatric Center - Texas Medical Center, Houston, Texas
  - University of Utah - PPDS, Salt Lake City, Utah
- Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- Croatia (2):
  - Klinika Za Djecje Bolesti Zagreb, Zagreb
  - University Hospital for Infection Diseases "Dr. Fran Mihaljevic" - PPDS, Zagreb
- France (3):
  - CHRU Montpellier; SMPEA Peyre Plantade Centre de Ressources Autisme, Montpellier
  - Hospital Necker, Paris
  - Assistance Publique Hopitaux de Paris, Val-de-Marne
- Germany (2):
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Ulm, Ulm
- Hippokration Hospital, Thessaloniki, Greece
- Italy (2):
  - IRCCS Ospedale Pediatrico Bambino Gesù - INCIPIT - PIN, Rome, Lazio
  - ASST di Lecco - Presidio Ospedaliero A. Manzoni di Lecco, Lecco, Lombardy
- Szpital Kliniczny im Karola Jonschera Uniwersytetu Medycznego im Karola Marcinkowskiego w Poznaniu, Poznan, Poland
- Global Clinical Trials Sunnyside, Pretoria, South Africa
- Spain (4):
  - Hospital Sant Joan de Deu - PIN; Unitat de Recerca - Farmacia, Esplugues de Llobregat, Barcelona
  - Hospital Infantil Universitario Niño Jesus; Sección de Neuropediatria, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
- Great North Childrens Hospital, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).